CLINICAL TRIAL: NCT01941914
Title: Calcium Electroporation for the Treatment of Keloids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Julie Gehl, Medical doctor, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA1310
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Keloid
Keywords: Calcium electroporation; calcium; electroporation; electrotransfer; keloid
MeSH Terms: conditions — Keloid | interventions — Calcium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcium electroporation (Experimental): The keloid will be treated with intratumoral injection of calcium chloride followed by electrotransfer. It is a once only treatment.
  Calcium chlorid concentration is 9 mg/ml Total dose is 0,5ml/cm3 tumor volume.
  Interventions: Drug: Calcium chloride

INTERVENTIONS:
Drug: Calcium chloride
  Other Names: Calcium Chloride dihydrate; ATC code A02AC; EV substance codeSUB12664MIG

SUMMARY:
The purpose of this study is to evaluate the effect of calcium electroporation on keloids.

DETAILED DESCRIPTION:
The keloids wil be treated with intratumoral injection of calcium followed by electroporation. It is a once only treatment and the patients will be followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 keloid available to electroporation.
* Patient should have been offered standard treatment.
* At least 8 weeks since other keloid treatment.
* Performance status <2 (ECOG).
* Platelet count >50 mia/l
* International Normalized Ratio (INR) <1,2.
* Age >18.
* Patient should be able to understand participants information.
* Signed, informed consent.

Exclusion Criteria:

* Clinically significant coagulopathy.
* Pregnancy or lactation.
* Participation in other clinical trial involving experimental drugs or participation in a clinical trial within 4 weeks before study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Response evaluated by Vancouver Scar Scale | After 6 months
  Vancouver scar scale evaluate the keloids by: pigmentation, pliability, height, and vascularity.

SECONDARY OUTCOMES:
Adverse events to calcium electroporation. | After 6 months.
  Describe adverse events using Common Terminology for Adverse Events, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Oncology, Copenhagen University hospital, Herlev, Herlev, Denmark